CLINICAL TRIAL: NCT03101059
Title: Evaluation of the Presence of Airway Collapse in Patients With Mounier-Kuhn Syndrome and Titration With Continuous Positive Pressure Through Non-invasive Mechanical Ventilation to Reduce Collapse
Brief Title: Airway Collapse in Patients With Mounier-Kuhn Syndrome: Titration With Positive Pressure to Reduce Collapse
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Principal Investigator, Rafael Stelmach, Clinical Professor, University of Sao Paulo General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: CAAE64001317400000068
Record Dates: First submitted 2017-03-23; First posted 2017-04-04 (Actual); Last update posted 2017-10-26 (Actual); Status verified 2017-10

CONDITIONS: Mounier-Kuhn Syndrome
Keywords: Tracheal; Bronchial; Tracheobronchiomegaly; Collapse; obstructive sleep apnea syndrome; Computer Tomography; Impedance Tomography
MeSH Terms: conditions — Tracheobronchomegaly; Unconsciousness; Sleep Apnea, Obstructive

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MKS pax (Experimental): Munier-Kuhn Syndrome patients
  Interventions: Procedure: Non invasive ventilation - Continuous Positive Airway Pressure

INTERVENTIONS:
Procedure: Non invasive ventilation - Continuous Positive Airway Pressure — To identify, through bronchoscopy, the prevalence of collapse and whether it is possible to counteract an optimum pressure generated by NIV with CPAP that reduces tracheal and bronchial collapse in patients with SMK; To study the frequency of OSAS in patients with MKS ; Record reversal of collapse with CPAP using chest tomography; To identify the impact of CPAP on the distribution of pulmonary ventilation through the analysis of electrical impedance tomography.

SUMMARY:
Mounier-Kuhn syndrome (MKS), or congenital tracheobronchiomegaly, is an entity characterized by dilation of the trachea and bronchi, associated with respiratory infections.The main signs and symptoms are cough, bulging and purulent expectoration, digital clubbing, dyspnoea, and wheezing.Some of these symptoms are believed to be due to excessive collapse of the intra-thoracic trachea and bronchi, resulting in airways obstruction of more than 50% . The purpose of this study is to identify and reduce tracheal collapse.

DETAILED DESCRIPTION:
Mounier-Kuhn syndrome (MKS), or congenital tracheobronchiomegaly, is an entity characterized by dilation of the trachea and bronchi, associated with respiratory infections. The prevalence among patients with respiratory symptoms is 0.4 to 1.6%. Its histological features include the atrophy or absence of longitudinal elastic fibers and smooth muscle cells of the airways, responsible for the structural alterations found, such as tracheobronchiomegaly, the presence of inter cartilaginous diverticula, bulging and dilation of the walls of the trachea and bronchi. The main signs and symptoms are cough, bulging and purulent expectoration, digital clubbing, dyspnoea, and wheezing and wheezing accompanied by recurrent respiratory infection. There may be association with other comorbidities such as gastroesophageal reflux disease, chronic obstructive pulmonary disease, bronchiectasis and obstructive sleep apnea / hypopnea syndrome (OSAS). Some of these symptoms are believed to be due to the tracheobronchial disease present in some patients, defined by excessive collapse of the intrathoracic trachea and bronchi resulting in airways obstruction of more than 50%. The main clinical impact is obstruction to expiratory airflow, with consequent air entrapment, reduction of cough and bronchial hygiene effectiveness, facilitating recurrent respiratory infections. Because it is a rare morbidity and little studied, the specific therapy is not consensual, and the main interventions are extrapolated from other pathologies. The use of non invasive mechanical ventilation (NIMV) with continuous positive airway pressure (CPAP) is reported as an option for treatment, however, there are no randomized studies proving its efficacy. The purpose of this study is to identify and reduce tracheal collapse and bronchi of SMK carriers with the use of positive pressure (CPAP-NIV) and to analyse their repercussion in the small airways.

ELIGIBILITY:
Inclusion Criteria:

* Has Mounier-Khun Syndrome
* Accept and signed informed consent form

Exclusion Criteria:

* Other morbidity avoiding study procedures

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2017-06-08 (Actual); Primary Completion 2018-09 (Estimated); Study Completion 2019-04 (Estimated)

PRIMARY OUTCOMES:
Percentage of tracheal-bronchial collapse area before and after applied positive pressure through bronchoscopy | 18 months
  Identify the prevalence of collapse and whether it is possible to counteract an optimum pressure generated by NIV with CPAP that reduces tracheal and bronchial collapse in patients with SMK

SECONDARY OUTCOMES:
Apnea+hypopnea (AHI) index in patients with SMK | 24 months
  Study the frequency of OSAHS in patients with SMK;
Percentage of tracheal-bronchial collapse area before and after applied positive pressure measure using chest tomography | 24 months
  Record reversal of collapse with CPAP using chest tomography
Inspiratory and expiratory lung volumes before and after applied positive pressure measure using electrical impedance tomography. | 24 months
  To identify the impact of CPAP on the distribution of pulmonary ventilation through the analysis of electrical impedance tomography.

CONTACTS AND LOCATIONS:
Locations (1):
- Divisao de Pneumologia, Instituto do Coracao, Hospital das Clinicas HCFMUSP, Faculdade de Medicina, Universidade de Sao Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lima E, Nakamura MAM, Genta PR, Rodrigues AJ, Athanazio RA, Rached S, Costa ELV, Stelmach R. Improving Airways Patency and Ventilation Through Optimal Positive Pressure Identified by Noninvasive Mechanical Ventilation Titration in Mounier-Kuhn Syndrome: Protocol for an Interventional, Open-Label, Single-Arm Clinical Trial. JMIR Res Protoc. 2020 Aug 14;9(8):e14786. doi: 10.2196/14786. PMID 32795996